CLINICAL TRIAL: NCT07226999
Title: A GLOBAL PHASE 2/3 INTERVENTIONAL STUDY OF PF-08634404 IN COMBINATION WITH CHEMOTHERAPY IN PARTICIPANTS WITH EXTENSIVE STAGE SMALL CELL LUNG CANCER
Brief Title: A Study to Learn About the Study Medicine Called PF-08634404 in Combination With Chemotherapy in Adult Participants With Extensive-Stage Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C6461004; 2025-523522-41-00 (EU CTIS Number); Symbiotic-Lung-04 (Other: Pfizer)
Record Dates: First submitted 2025-11-07; First posted 2025-11-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Small Cell Lung Cancer (SCLC)
Keywords: small cell lung cancer; extensive stage small cell lung cancer; first-line
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Phase 2 is open-label, whereas Phase 3 is double-blind, randomized design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 2 Single arm (Experimental): Participants will receive PF-08634404 in combination with chemotherapy
  Interventions: Drug: PF-08634404; Drug: Chemotherapy
- Phase 3 Experimental Arm (Experimental): Participants will receive PF-08634404 in combination with chemotherapy
  Interventions: Drug: PF-08634404; Drug: Chemotherapy
- Phase3 Control Arm (Active Comparator): Participants will receive atezolizumab in combination with chemotherapy
  Interventions: Biological: Atezolizumab; Drug: Chemotherapy

INTERVENTIONS:
Drug: PF-08634404 — Concentrate for solution for infusion
  Arms: Phase 2 Single arm; Phase 3 Experimental Arm
Biological: Atezolizumab — Injection for intravenous use
  Arms: Phase3 Control Arm
Drug: Chemotherapy — Injection for intravenous use

SUMMARY:
This study is being done to learn more about a new medicine called PF-08634404 and how well it works when given with chemotherapy to adults with extensive-stage small cell lung cancer (ES-SCLC), a fast-growing type of lung cancer that has spread widely in the body.

To join the study, participants must meet the following conditions:

* Be 18 years or older.
* Have extensive-stage small cell lung cancer confirmed by lab tests.
* Have not received chemotherapy or radiation for this type of lung cancer.
* Be in good physical condition and have healthy organs based on medical tests.

The study has two parts:

* In the first part, researchers will check how safe the study medicine is and how well people tolerate it when given with chemotherapy.
* In the second part, they will compare study medicine plus chemotherapy to another approved treatment (atezolizumab plus chemotherapy) to see which works better.

Participants will receive the treatment through IV infusions (medicine given directly into a vein). The treatment will be given in repeated time periods called cycles. Some participants will continue receiving the study medicine alone after the initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed extensive-stage small cell lung cancer (ES-SCLC).
* Participants have not received systemic therapy (chemotherapy, radiotherapy, chemoradiation) for ES-SCLC.
* Treatment-free for at least 6 months since last chemo/radiotherapy, among those treated (with curative intent) with prior chemo/radiotherapy for limited-stage SCLC
* Have at least one measurable lesion as the targeted lesion based on RECIST V1.1.
* Eastern Cooperative Oncology Group performance status of 0 or 1.
* Adequate organ function

Exclusion Criteria:

* known active CNS lesions, including brainstem, meningeal, or spinal cord metastases or compression
* Leptomeningeal disease
* Clinically significant risk of hemorrhage or fistula
* history of another malignancy within 3 years
* active autoimmune diseases requiring systemic treatment within the past 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-12-09 (Actual); Primary Completion 2030-06-14 (Estimated); Study Completion 2034-03-11 (Estimated)

PRIMARY OUTCOMES:
Phase 2: Confirmed Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1] based on the investigator's assessment | Up to approximately 2 years after completion of study treatment of last study participant
  Defined as the proportion of participants in whom a confirmed complete response (CR) or partial response (PR) is observed as best overall response. ORR using RECIST v1.1 as assessed by investigator.
Phase 2: Number of participants with treatment-emergent adverse events | Up to 90 days after the last dose of treatment
  Adverse Events (AEs) as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), timing, seriousness, and relationship to study intervention.
Phase 3: Overall Survival (OS) | Up to approximately 2 years after completion of study treatment of last study participant
  OS is defined as the time from the date of randomization to the date of death due to any cause. OS is secondary outcome measure in Phase 2 portion of the study.

SECONDARY OUTCOMES:
Duration of Response (DOR) as assessed by Investigator based on RECIST v1.1 | Up to approximately 2 years after completion of study treatment of last study participant
  DOR is defined as the time from the first documentation of objective response (CR or PR) to the date of first documentation of PD or death due to any cause.
Progression Free Survival (PFS) as assessed by investigator based on RECIST v1.1 | Up to approximately 2 years after completion of study treatment of last study participant
  PFS is defined as the time from the date of randomization to the date of first documented disease progression, per RECIST v1.1, or death to any cause, whichever occurs first
Number of participants with Laboratory abnormalities | Up to 90 days after the last dose of treatment
  Laboratory abnormalities as characterized by type, frequency, severity (as graded by NCI CTCAE version 5.0), and timing.
Phase 2: Number of Participants who Experience a Dose-Limiting Toxicity (DLT) | Up to 90 days after the last dose of treatment
  DLT (any of the prespecified AEs that are attributable to study treatment(s), excluding toxicities clearly due to underlying disease or extraneous causes) rate estimated based on data from DLT-evaluable participants during the DLT evaluation period.
Pharmacokinetics: Serum concentrations of PF-08634404 | Up to 37 days after the last dose of treatment
Incidence of antidrug antibody against PF-08634404 | Up to 37 days after the last dose of treatment
Phase 2: Overall Survival | Up to approximately 2 years after completion of study treatment of last study participant
  Overall survival defined as the time from the date of randomization to the date of death due to any cause.
Phase 3: PFS using RECIST v1.1 as assessed by blinded independent central review (BICR) | Up to approximately 2 years after completion of study treatment of last study participant
  Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of the first documentation of objective progressive disease (PD) assessed by BICR per RECIST v1.1, or death due to any cause, whichever occurs first.
Phase 3: Confirmed ORR using RECIST v1.1 as assessed by BICR | Up to approximately 2 years after completion of study treatment of last study participant
  ORR is defined as the proportion of participants in the analysis population having a best overall response (BOR) of confirmed CR or confirmed PR according to RECIST v1.1 as assessed by BICR.
Phase 3: DOR using RECIST v1.1 as assessed by BICR | Up to approximately 2 years after completion of study treatment of last study participant
  The time from the first documentation of objective response (CR or PR that is subsequently confirmed) to the date of the first documentation of PD as determined by BICR assessment per RECIST v1.1, or death due to any cause, whichever occurs first.
Phase 3: Mean scores and Change from baseline in the global health status/quality of life (QoL), function, and symptom scores on the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Up to approximately 2 years after completion of study treatment of last study participant
  The EORTC QLQ-C30 is a questionnaire for quantitative measure of health-related quality of life pertinent to participants with a broad range of cancers who are participating in international clinical trials.
Phase 3: Mean scores and Change from Baseline on the EORTC Quality of Life Cancer Questionnaire - Lung Cancer 13 (EORTC QLQ-LC13) | Up to approximately 2 years after completion of study treatment of last study participant
  EORTC QLQ-LC13 is a lung cancer specific module that serves as an additional 13 item questionnaire to the general EORTC cancer questionnaire, the EORTC QLQ-C30.
Phase 3: Time to definitive deterioration (TTdD) in the global health status/QoL, function, and symptom scores on the EORTC QLQ-C30 | Up to approximately 2 years after completion of study treatment of last study participant
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.
Phase 3: TTdD in the dyspnea, cough, and chest pain scores on the EORTC QLQ-LC13 | Up to approximately 2 years after completion of study treatment of last study participant
  TTdD is defined as the time from date of randomization to first onset of Patient Reported Outcome (PRO) deterioration without subsequent recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (4):
  - Highlands Oncology Group, Springdale, Arkansas
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - Gulf Coast, Webster, Texas
- Kansai Medical University Hospital, Hirakata, Osaka, Japan
- Pan American Center for Oncology Trials, LLC, San Juan, Other, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests